CLINICAL TRIAL: NCT06381011
Title: Can Local Vibration be Used to Alleviate Symptoms of Cervical Radiculopathy?
Brief Title: Local Vibration in Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEUFTR-4
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cervical Radiculopathy
Keywords: neck pain; paresthesia
MeSH Terms: conditions — Radiculopathy; Neck Pain; Paresthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The evaluator and the researcher administering the local vibration application will be different. Patients will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Local Vibration Group (Sham Comparator): In addition to conventional treatment program the placebo local vibration application will be applied bilaterally to the cervicothoracic region of the patients in the placebo group. For the application, the patient will be placed in an upright sitting position, and the local vibration device will be moved without touching the patient's skin while it is operational.
  Interventions: Other: Local Vibration
- Local Vibration Intervention Group (Experimental): In addition to conventional treatment program the patients in this group will receive bilateral local vibration application on the cervicothoracic region, utilizing two different frequency values, 50 Hz and 100 Hz. Initially, a flat attachment will be placed on the device, and application will be performed on the neck and back regions for 5 minutes at a frequency of 50 Hz. Then, the other attachment of the device will be used, the frequency value will be increased to 100 Hz, and application will be performed on a total of 5 sensitive points specified by the manufacturer in the neck and back regions, with one minute per point for a total of 5 minutes. Local vibration will be applied to each side for ten minutes, totaling 20 minutes, and this will be conducted for five consecutive days. To determine which side to start the application from, a coin toss will be performed.
  Interventions: Other: Local Vibration

INTERVENTIONS:
Other: Local Vibration — The patients in the study group will receive local vibration application including different frequency values on the neck and back regions for five consecutive days.

SUMMARY:
The aim of this study is to evaluate the effect of local vibration application on the upper extremity pain, paresthesia, neck pain, and limitations in cervical joint range of motion experienced by patients with cervical radiculopathy.

DETAILED DESCRIPTION:
At least 34 patients diagnosed with cervical radiculopathy who meet the inclusion and exclusion criteria will be included in the study. Subsequently, the patients will be randomly divided into two groups. Patients in the first group will receive placebo local vibration application in addition to conventional treatment, while patients in the second group will receive local vibration application in addition to conventional treatment

ELIGIBILITY:
Inclusion Criteria:

* 1. Between the ages of 18 and 70,
* 2. Nerve root compression according to the magnetic resonance imaging,
* 3. Unilateral or bilateral neck pain rated 3 or higher on the Numeric Pain Rating Scale, or neck pain with paresthesia or upper extremity pain rated 3 or higher on the Numeric Pain Rating Scale.

Exclusion Criteria:

* 1. History of previous cervical or thoracic spinal surgery,
* 2. Symptoms or signs of upper motor neuron disorder,
* 3. Body mass index (BMI) higher than 35 kg/m2,
* 4. Having received spinal injection in the last two weeks,
* 5. Presence of local infection at the application site,
* 6. Upper extremity nerve entrapment syndrome (such as carpal tunnel or cubital tunnel syndrome),
* 7. Diagnosis of systemic inflammatory arthritis (such as rheumatoid arthritis, etc.),
* 8. Having engaged in strenuous exercise in the last 24 hours,
* 9. Poor or noncompliance to the treatment program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Neck Pain | Change from baseline neck pain immediately and five days after the intervention
  The effect of local vibration intervention on patients' neck pain will be evaluated using the Patients' Global Impression of Improvement Scale. In this scale, patients will be asked to mark their perceived change in pain using the following options: 'very much better,' 'much better,' 'a little better,' 'no change,' 'a little worse,' 'much worse,' and 'very much worse.'
Upper Limb Pain | Change from baseline neck pain immediately and five days after the intervention
  The effect of local vibration intervention on patients' upper limb pain will be evaluated using the Patients' Global Impression of Improvement Scale. In this scale, patients will be asked to mark their perceived change in pain using the following options: 'very much better,' 'much better,' 'a little better,' 'no change,' 'a little worse,' 'much worse,' and 'very much worse.'
Paresthesia | Change from baseline neck pain immediately and five days after the intervention
  The effect of local vibration intervention on patients' paresthesia will be evaluated using the Patients' Global Impression of Improvement Scale. In this scale, patients will be asked to mark their perceived change in paresthesia using the following options: 'very much better,' 'much better,' 'a little better,' 'no change,' 'a little worse,' 'much worse,' and 'very much worse.'

SECONDARY OUTCOMES:
Cervical Range of Motion | Change from baseline neck pain immediately and five days after the intervention
  The immediate and short-term effect of local vibration intervention on cervical range of motion will be measured using a 10-inch standard manual goniometer. To measure cervical flexion and extension range of motion, the pivot point of the goniometer will be placed at the external auditory meatus. The fixed arm of the goniometer will be held vertically, and the moving arm will follow along the base of the nostrils. For measuring cervical rotation range of motion, measurements will be taken from behind the participants. The pivot point of the goniometer will be placed at the vertex, while the fixed arm will be kept parallel to the acromion, and the moving arm will follow along with their nose. Lateral flexion range of motion will be taken in front of the participants. The pivot point of the goniometer will be placed over the sternal notch, with its fixed arm parallel to the acromion, and its moving arm will follow along the tip of the participants' nose.
The Change in the Pressure Pain Threshold of the Upper Trapezius | Change from baseline neck pain immediately and five days after the intervention
  The potential impact of local vibration intervention on patients' pain thresholds will be evaluated using an analog algometer. Pain threshold measurements will be taken at the upper trapezius muscle. The algometer will be positioned perpendicular to the measurement areas. Three measurements will be taken for each region, with a half-minute interval between measurements. The average of the three measurements will be calculated and recorded. A change of 20-25% in the algometric measurement values will be considered significant.
The Change in the Viscoelastic Properties of the Upper Trapezius | Change from baseline neck pain immediately and five days after the intervention
  The effect of local vibration intervention on the viscoelastic properties of patients' upper trapezius will be measured using the myotonometer (MyotonPRO). The upper trapezius myometric measurement will be taken with the patient seated on a chair with hands placed over knees, and measured from the midpoint between the C7 spinous process and the acromion.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; Gökmen Reyhanlı, M.D., Principal Investigator — Bitlis Tatvan State Hospital; Erhan Dincer, M.Sc., Principal Investigator — Bitlis Eren University; Abdurrahman Tanhan, Ph.D., Principal Investigator — Bitlis Eren University; Etem Öztürk, Principal Investigator — Bitlis Tatvan State Hospital
Locations (1):
- Bitlis Tatvan State Hospital, Bitlis, Tatvan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wainner RS, Fritz JM, Irrgang JJ, Boninger ML, Delitto A, Allison S. Reliability and diagnostic accuracy of the clinical examination and patient self-report measures for cervical radiculopathy. Spine (Phila Pa 1976). 2003 Jan 1;28(1):52-62. doi: 10.1097/00007632-200301010-00014. PMID 12544957
- [Background] Young IA, Michener LA, Cleland JA, Aguilera AJ, Snyder AR. Manual therapy, exercise, and traction for patients with cervical radiculopathy: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):632-42. doi: 10.2522/ptj.20080283. Epub 2009 May 21. PMID 19465371
- [Background] Thoomes EJ, van Geest S, van der Windt DA, Falla D, Verhagen AP, Koes BW, Thoomes-de Graaf M, Kuijper B, Scholten-Peeters WGM, Vleggeert-Lankamp CL. Value of physical tests in diagnosing cervical radiculopathy: a systematic review. Spine J. 2018 Jan;18(1):179-189. doi: 10.1016/j.spinee.2017.08.241. Epub 2017 Aug 31. PMID 28838857
- [Background] Wong JJ, Cote P, Quesnele JJ, Stern PJ, Mior SA. The course and prognostic factors of symptomatic cervical disc herniation with radiculopathy: a systematic review of the literature. Spine J. 2014 Aug 1;14(8):1781-9. doi: 10.1016/j.spinee.2014.02.032. Epub 2014 Mar 12. PMID 24614255
- [Background] Young IA, Pozzi F, Dunning J, Linkonis R, Michener LA. Immediate and Short-term Effects of Thoracic Spine Manipulation in Patients With Cervical Radiculopathy: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2019 May;49(5):299-309. doi: 10.2519/jospt.2019.8150. Epub 2019 Apr 25. PMID 31021691
- [Background] Ayub A, Osama M, Ahmad S. Effects of active versus passive upper extremity neural mobilization combined with mechanical traction and joint mobilization in females with cervical radiculopathy: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(5):725-730. doi: 10.3233/BMR-170887. PMID 30664500
- [Background] Rubinstein SM, Pool JJ, van Tulder MW, Riphagen II, de Vet HC. A systematic review of the diagnostic accuracy of provocative tests of the neck for diagnosing cervical radiculopathy. Eur Spine J. 2007 Mar;16(3):307-19. doi: 10.1007/s00586-006-0225-6. Epub 2006 Sep 30. PMID 17013656
- [Background] Taso M, Sommernes JH, Kolstad F, Sundseth J, Bjorland S, Pripp AH, Zwart JA, Brox JI. A randomised controlled trial comparing the effectiveness of surgical and nonsurgical treatment for cervical radiculopathy. BMC Musculoskelet Disord. 2020 Mar 16;21(1):171. doi: 10.1186/s12891-020-3188-6. PMID 32178655
- [Background] Alshami AM, Bamhair DA. Effect of manual therapy with exercise in patients with chronic cervical radiculopathy: a randomized clinical trial. Trials. 2021 Oct 18;22(1):716. doi: 10.1186/s13063-021-05690-y. PMID 34663421
- [Background] Abbed KM, Coumans JV. Cervical radiculopathy: pathophysiology, presentation, and clinical evaluation. Neurosurgery. 2007 Jan;60(1 Supp1 1):S28-34. doi: 10.1227/01.NEU.0000249223.51871.C2. PMID 17204882